CLINICAL TRIAL: NCT03403894
Title: Description of Practices Implemented in the Birth of Living Children Before 24 Weeks of Amenorrhea
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 17-AOI-01
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Infant, Extremely Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Asking caregivers in their practice — A questionary is given to caregivers

SUMMARY:
Every year, at the Nice University Hospital, about sixty deliveries take place before 24 weeks of amenorrhea. The child is not viable because of his extreme immaturity. In most cases, a child born before 24 years of age is stillborn, but in about one in three cases, it shows signs of life such as heartbeat, breathing, gasps or limb movements.

With these too small children showing signs of life, three attitudes are possible: doing nothing and waiting for this life to stop by themselves, setting up palliative care to ensure the child's comfort, or administering a medication to shorten his or her life. The attitude to have is not univocal and the feeling of the teams confronted with their management is difficult even if the goal of the caregivers is always to act as best as possible.

The main objective of the study is to describe the clinical state of the child and the practices implemented in the birth room at the Nice University Hospital when children showing signs of life before 24 weeks of amenorrhea are born.

The secondary objective is to describe caregivers' experiences, their experiences of these situations and attitudes towards children and their parents, and to identify ethical dilemmas in these situations.

This study is an observational cohort study including all births of live children before 24 weeks of amenorrhea at Nice University Hospital for 12 months. It consists of two parts: a quantitative study describing the child's condition and caregiving practices, and a qualitative study of caregivers' experiences and the determinants of their attitudes towards the child.

The investigator will coordinate the collection of the data necessary to conduct the quantitative study, and then conduct individual semi-directive interviews with each of the caregivers present at the birth of the child. The qualitative study will be based on the analysis of these interviews.

ELIGIBILITY:
Inclusion Criteria:

* Child born before 24 weeks of amenorrhea (term estimated by echographic dating or by the date of the last menstrual period in the absence of ultrasound)
* Inscription in the birth register (so from 15 weeks of amenorrhea)
* Non-opposition of the parents

Exclusion Criteria:

- Child transferred to neonatal intensive care unit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Child born before 24 weeks of amenorrhea will be study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Existence of cardiac activity | 5 hours
Presence of respiratory movements and/or gasps | 5 hours
Existence of limb movements | 5 hours
Place of care | 5 hours
Identification of the function of the caregiver(s) who performed the care | 5 hours
Conditions of installation of the child (position, skin-to-skin...) | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Céline MARTIN, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No